CLINICAL TRIAL: NCT05304429
Title: Application of a Nutritional Counseling Program on the Frailty of Older Adults in the Mexican Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Principal Investigator, Mariana Cecilia Orellana Haro, Clinical Proffessor, Instituto Tecnologico y de Estudios Superiores de Monterey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMAZGA-APPR.001
Record Dates: First submitted 2022-03-08; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Frailty Syndrome
MeSH Terms: conditions — Frailty | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Clinical trial with intervention group and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nutritional counseling group (Experimental): This group will have nutrition education sessions every fifteen days and will keep track of 10 healthy behaviors through goal setting and self-monitoring.
  Interventions: Behavioral: nutrition education; Behavioral: nutritional counseling
- group without nutritional counseling (No Intervention): This group will have sessions every fifteen days of reading, knitting and other activities unrelated to health.

INTERVENTIONS:
Behavioral: nutrition education — Educational sessions with topics that will address the management and prevention of frailty syndrome focusing on protein intake and physical activity
  Arms: nutritional counseling group
Behavioral: nutritional counseling — nutritional counseling system based on the com-b model through three strategies: goal setting, self-monitoring and social support
  Arms: nutritional counseling group

SUMMARY:
In the present study, the COM-B model is intended to be used as a central axis in the planning of the nutritional counseling intervention, since it proposes that behavioral modification is conditioned by the capacity, opportunity and motivation of the person, 3 basic components that can be addressed with nutritional education and goal-setting strategies, self-monitoring and social support.

The intervention will consist of applying nutritional counseling in older adults with frailty syndrome to measure the effect on indicators of this syndrome such as nutritional status, handgrip strength, protein consumption and physical activity.

DETAILED DESCRIPTION:
Clinical trial with intervention group and control group that include men and women over 60 years of age with frailty or risk of suffering it according to the frailty scale

INTERVENTION:

The COM-B system is based on 3 main pillars that appear in the initials of its name, being the C for "capacity", the O for "opportunity" and the M for "motivation". The behavior of the person is attributed to these in such a way that if they have the capacity, motivation and opportunity, the strategies used for behavior change will be more effective.

Based on this theory, the investigators support the intervention of the study in which the capacity of the participants will be developed through nutritional education, motivation through goal setting and self-monitoring, and the opportunity for social support that will be provided through this project at no cost to users of the DIF Zapopan Metropolitan Center for the Elderly.

Regarding the establishment of goals, 10 important behaviors will be worked on to prevent or combat frailty, which promote adequate protein consumption, balance in the distribution of nutrients, avoid prolonged periods of fasting by encouraging the consumption of healthy snacks, decreased consumption of ultra-processed foods, increasing the consumption of plant-based foods and performing strength exercises. The adherence to these behaviors will be self-monitored on a weekly basis through a format (see annex 4) that each person will receive and that is inspired by the strategy used by Beeken and collaborators in the "ten top tis" project where the effectiveness in behavioral modification through goal setting and self-monitoring.

Nutritional education was carried out in group sessions of 40 minutes having a total of 10 workshops which provided practical theoretical tools to each of the behaviors to be monitored, in this way each workshop addressed a specific behavior.

The intervention will be aimed at qualitatively and quantitatively modifying eating habits, emphasizing protein consumption and modifying physical activity habits, limiting sedentary behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 60 years of age
* That they have a normal cognitive function (more than 24 points in the minimental test)
* That they attend weekly the Metropolitan Center for the Elderly (DIF Zapopan)
* Who suffer from frailty or pre-frailty (from 1 to 5 points on the frailty scale)

Exclusion Criteria:

* Severe dysphagia
* Consumption of food supplements (protein powder or vitamins)
* Senile dementia, cognitive impairment or Alzheimer's
* People who are following a diet or physical activity plan prescribed by a professional

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-29 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Frailty syndrome | 6 months
  Geriatric syndrome characterized by a decreased ability of the body to respond to external stressors, causing in the individual: risk of falls, functional decline, disability, dependency, institutionalization and even death.
  For its evaluation, the frailty scale valid in Mexicans proposed by Díaz de León González in 2016 will be used.
  It considers 5 questions and classifies those with a score between 3 to 5 points as frail, pre-fragile between 1 and 2 and non-fragile with a score of zero.
  Questions:
  Do you feel tired most of the time? Can you walk up one flight of stairs without breaks or help? Are you able to walk 100 m without pausing and without assistance? Have more than 5 symptoms. Arthritis, diabetes, angina/heart attack, hypertension, stroke, asthma, chronic bronchitis, emphysema, osteoporosis, colorectal cancer, skin cancer, depression/anxiety, dementia, leg ulcers.
  Weightloss: > 5% in the last year

SECONDARY OUTCOMES:
Protein intake | 6 months
  Intake of grams of protein per day from animal or vegetable sources. It will be evaluated through a 24-hour recall.
Malnutrition | 6 months
  Malnutrition is a lack of calories or one or more essential nutrients. It will be measured through the Mini Nutritional Assessment long form (MNA-LF), a screening tool to help identify elderly patients who are malnourished or at risk of malnutrition.
  The tool consists of a 18-item in the long form scale.
Handgrip strength | 6 months
  It is the maximum isometric strength of the hand and forearm muscles.. It will be evaluated through the pressure force of the participant's dominant hand estimated through a dynamometer and whose cut-off points refer to a decrease in force when it is below 30 kg in men or 20 kg in women.
sedentary activities | 6 months
  Those activities that people do sitting or reclining, while we are awake, and that use very little energy.
  These will be evaluated through self-report of sedentary activities Adapted from the ASAQ Questionnaire (Adolescent Sedentary Activity Questionnaire)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nykanen I, Rissanen TH, Sulkava R, Hartikainen S. Effects of individual dietary counseling as part of a comprehensive geriatric assessment (CGA) on nutritional status: a population-based intervention study. J Nutr Health Aging. 2014 Jan;18(1):54-8. doi: 10.1007/s12603-013-0342-y. PMID 24402390
- [Background] Andersson J, Hulander E, Rothenberg E, Iversen PO. Effect on Body Weight, Quality of Life and Appetite Following Individualized, Nutritional Counselling to Home-Living Elderly after Rehabilitation - An Open Randomized Trial. J Nutr Health Aging. 2017;21(7):811-818. doi: 10.1007/s12603-016-0825-8. PMID 28717811
- [Background] Faber MJ, Bosscher RJ, Chin A Paw MJ, van Wieringen PC. Effects of exercise programs on falls and mobility in frail and pre-frail older adults: A multicenter randomized controlled trial. Arch Phys Med Rehabil. 2006 Jul;87(7):885-96. doi: 10.1016/j.apmr.2006.04.005. PMID 16813773
- [Background] Gardner B, Jovicic A, Belk C, Kharicha K, Iliffe S, Manthorpe J, Goodman C, Drennan VM, Walters K. Specifying the content of home-based health behaviour change interventions for older people with frailty or at risk of frailty: an exploratory systematic review. BMJ Open. 2017 Feb 9;7(2):e014127. doi: 10.1136/bmjopen-2016-014127. PMID 28183809
- [Background] Fernandez-Barres S, Garcia-Barco M, Basora J, Martinez T, Pedret R, Arija V; Project ATDOM-NUT group. The efficacy of a nutrition education intervention to prevent risk of malnutrition for dependent elderly patients receiving Home Care: A randomized controlled trial. Int J Nurs Stud. 2017 May;70:131-141. doi: 10.1016/j.ijnurstu.2017.02.020. Epub 2017 Feb 23. PMID 28273591
- See also: findings of the national study of health and aging in Mexico — http://www.enasem.org/images/MHASFactSheet_Frailty_SPANISH.pdf